CLINICAL TRIAL: NCT01172691
Title: Randomized, Blinded, Controlled Trial of Inhaled Nitric Oxide (iNO) on Ischemia / Reperfusion Injury During Orthotopic Liver Transplantation With Marginal Grafts.
Brief Title: Trial of Inhaled Nitric Oxide (iNO) on Ischemia / Reperfusion Injury During Orthotopic Liver Transplantation With Marginal Grafts
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 010-085
Record Dates: First submitted 2010-07-28; First posted 2010-07-30 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Liver Transplant
Keywords: Liver transplant
MeSH Terms: interventions — Nitrogen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled Nitric Oxid (Experimental): iNO or placebo will be administered at 40 ppm during the procedure starting when the Warm Ischemia Time begins - liver from ice. Stop when patient transported to ICU
  Interventions: Drug: Inhaled Nitric Oxide (iNO)
- Placebo Arm (nitrogen) (Experimental): iNO or placebo will be administered at 40 ppm during the procedure starting when the Warm Ischemia Time begins - liver from ice. Stop when patient transported to ICU
  Interventions: Drug: Placebo Arm (Nitrogen)

INTERVENTIONS:
Drug: Inhaled Nitric Oxide (iNO) — iNO will be administered at 40 ppm during the procedure starting when the Warm Ischemia Time begins - liver from ice. Stop when patient transported to ICU
  Arms: Inhaled Nitric Oxid
Drug: Placebo Arm (Nitrogen) — Placebo will be administered at 40 ppm during the procedure starting when the Warm Ischemia Time begins - liver from ice. Stop when patient transported to ICU
  Arms: Placebo Arm (nitrogen)

SUMMARY:
This study is being done to determine if patients receiving (iNO) will have increased liver function and less damage from IR than patients who do not receive (iNO).

ELIGIBILITY:
Inclusion Criteria:

* Liver Transplant

Exclusion Criteria:

* Living donor transplants

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2014-01-22 (Actual)

PRIMARY OUTCOMES:
Evaluate the role of iNO in early ischemia reperfusion injury in marginal liver grafts during human orthotopic liver or liver/kidney transplantation. | 24 hours to 1 month

SECONDARY OUTCOMES:
iNO group will show accelerated restoration of liver allograft function following liver transplantation and this may translate to better clinical outcomes. Marginal grafts may function better in the treated group | 1 month to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Ramsay, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor Univsersity Medical Center, Dallas, Texas, United States